CLINICAL TRIAL: NCT02771132
Title: A Cluster-randomized Trial to Assess a Sexual Assault Prevention Intervention in Upper Primary School Adolescents in Nairobi, Kenya
Brief Title: A Cluster-randomized Trial to Assess a Sexual Assault Prevention Intervention in Adolescents in Nairobi, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: African Institute for Health and Development, Kenya (Unknown); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Mike Baiocchi, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34706
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Sexual Assault and Rape; Violence, Non-accidental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 12-hour intervention "IMPower" empowerment self defense course for girls and 12-hour Source of Strength for boys+ 2 refresher sessions (at 2 hrs. per session)
  Interventions: Behavioral: 12-hr "IMPower" empowerment self defense course; Behavioral: 12-hr Source of Strength for boys
- Standard of Care (Other): 1-2 hour course based on Ministry of Education life skills course (no refresher sessions)
  Interventions: Behavioral: Life-skills course

INTERVENTIONS:
Behavioral: 12-hr "IMPower" empowerment self defense course — The purpose of the 12-hr "IMPower" empowerment self defense course intervention for girls is to empower then to avoid risky situations, advocate for themselves, and, if needed, defend themselves against an attack.
  Arms: Intervention
Behavioral: 12-hr Source of Strength for boys — The 12-hr Source of Strength for boys curriculum is specifically designed for 10-13 year-old boys and focused on promoting gender equality, developing positive masculinity, and teaching safe and effective bystander intervention techniques.
  Arms: Intervention
Behavioral: Life-skills course — A 1.5-2 hour life skills class that is based on the Kenyan Ministry of Education life skills course and includes a wide range of topics, including sexual assault but also sanitation, food safety, and personal rights. All school-aged children who attend school typically receive this type of curriculum.
  Arms: Standard of Care

SUMMARY:
The primary objective of this study is to compare the effectiveness of classroom-based behavioral interventions (12-hour girls program and 12-hour boys program), to a standard-of care intervention, on reducing the incidence of self-reported sexual assault among girls from baseline.

Secondary objectives of this study is to determine the impact of the interventions on related physical and mental health status/outcomes, STI-risk behaviors, self-efficacy, and self-esteem.

DETAILED DESCRIPTION:
In Kenya, up to 46% of women report childhood sexual assault. In an implementation research project, a team at Stanford University will be pairing with three Kenyan NGO's to research the effectiveness of an intervention to prevent sexual assault among adolescent girls in the informal settlements around Nairobi, Kenya. The study design will be a cluster-randomized controlled trial with two arms comparing the intervention to a standard of care group. The intervention consists of two side-by-side behavioral and skills-based interventions, one for girls and one for boys, taught in schools. The interventions include identifying and avoiding risky situations, verbal techniques to diffuse situations, as well as bystander intervention techniques for boys and self-defense techniques for girls. Settlements with schools participating in the project include Kibera, Dandora, Huruma, and Mukuru.

This grant is part of the larger "What Works to Prevent Violence: A global program to prevent violence against women and girls" initiative, which is a large international initiative aimed at the prevention of gender-based violence. The initiative includes 18 projects from around the globe, and is supported by the Medical Research Council of South Africa, the London School of Hygiene and Tropical Medicine, and the UK Department for International Development (DFID). The primary contact people at Stanford University for this project are Clea Sarnquist, DrPH, MPH (cleas@stanford.edu) and Michael Baiocchi, PhD (baiocchi@stanford.edu).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 11-15 years
* Enrolled in the target schools
* Able to communicate in the study languages: English or Kiswahili

Exclusion Criteria:

* significant mental condition (learning difficulty, mental illness or substance abuse) which would impair their ability to consent to participation in the trial.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4121 (Actual)
Dates: Start 2015-09; Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Sexual Assault Incidence (WHO-Violence Against Women Survey) | 12 months
  self-reports of sexual assault within past 12 months, compared between control and intervention groups

SECONDARY OUTCOMES:
Physical Violence Incidence (WHO-Violence Against Women Survey) | 8-20 months post-intervention
  Self-reports of physical violence, compared between control and intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baiocchi, PhD, Principal Investigator — Stanford University
Locations (1):
- African Institute for Health and Development, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of the participants (who are minors), parties interested in the data should contact the investigators and provide evidence of IRB approval and data security safeguards at their institution(s). The sponsoring agency, DFID, anticipates making some of the data publicly available in the future.

REFERENCES:
- [Derived] Mphamba D, Solomon FR, Nyairo G, Kim CJ, Krishnamoorthi M, Edem B, Amuyunzu-Nyamongo M, Kang J, Baiocchi M, Sarnquist CC. Youth voices from an informal settlement of Nairobi, Kenya: Engaging adolescent perspectives on violence to inform prevention. Glob Public Health. 2022 Dec;17(12):3686-3699. doi: 10.1080/17441692.2022.2076895. Epub 2022 May 17. PMID 35579915
- [Derived] Sarnquist C, Kang JL, Amuyunzu-Nyamongo M, Oguda G, Otieno D, Mboya B, Omondi N, Kipkirui D, Baiocchi M. A protocol for a cluster-randomized controlled trial testing an empowerment intervention to prevent sexual assault in upper primary school adolescents in the informal settlements of Nairobi, Kenya. BMC Public Health. 2019 Jun 27;19(1):834. doi: 10.1186/s12889-019-7154-x. PMID 31248392
- See also: This protocol is part of the What Works to Prevent Violence Initiative, a global program to prevent violence against women and girls — http://www.whatworks.co.za/